CLINICAL TRIAL: NCT07233798
Title: Correlation of the Presence of Dural Pulsation With Clinical and Radiological Parameters in Patients Diagnosed With Lumbar Spinal Stenosis
Brief Title: Presence of Dural Pulsation in Patients Diagnosed With Lumbar Spinal Stenosis
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haner Direskeneli, Professor, Marmara University
Other Study IDs: MarmaraU-FTR-FBA-01
Record Dates: First submitted 2025-07-01; First posted 2025-11-18 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spinal Stenosis; Numerical Rating Scale; Disability Physical; Magnetic Resonance; Claudication
Keywords: Dural Pulsation; oswestry disability index
MeSH Terms: conditions — Spinal Stenosis; Intermittent Claudication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for dural pulsation
- Negative for dural pulsation

SUMMARY:
Lumbar spinal stenosis is defined as the narrowing of the spinal canal resulting from degenerative changes in the spinal joints, intervertebral discs, and the ligamentum flavum.

Pressure fluctuations within the cerebral and spinal vascular systems lead to the formation of pulsations. The periodic occurrence of these pulsations in the dura mater is referred to as spinal dural pulsation.The vibratory movements of the dura mater have been interpreted as an indicator that the spinal cord is freely mobile within the subarachnoid space and not subjected to any external compression.This study aims to investigate whether the presence of dural pulsation is associated with clinical and radiological parameters in patients diagnosed with lumbar spinal stenosis

DETAILED DESCRIPTION:
Lomber spinal stenosis is defined as a narrowing of the spinal canal resulting from degenerative changes in the spinal joints, intervertebral discs, and the ligamentum flavum. The reduction in the space surrounding the neurovascular structures may lead to significant clinical symptoms such as neurogenic claudication, radiating pain in the lower extremities, low back pain, and urinary or fecal incontinence. Symptoms often improve when patients sit down or lean forward. However, if the pain induced by standing or walking postures becomes severe, it may impair the ability to perform daily and independent activities.

Magnetic Resonance Imaging is the primary imaging modality for the diagnosis of LSS. It provides high sensitivity and specificity in identifying anatomical abnormalities such as disc herniation, facet joint degeneration, and hypertrophy of the ligamentum flavum. However, as MRI findings may be influenced by factors such as patient positioning and imaging protocols, the interpretation of MRI should always be correlated with clinical findings in the diagnosis of LSS.

Periodic oscillations within the central nervous system occur due to pressure changes in the cerebral and spinal vascular systems. The rhythmic occurrence of these oscillations at the level of the dura mater is referred to as spinal dural pulsation. In previous studies, the vibratory movements of the spinal cord, dura mater, and cerebrospinal fluid (CSF) have been observed intraoperatively and evaluated in detail using MRI. Surgeons have interpreted these rhythmic movements of the dura mater as an indication that the spinal cord is freely suspended within the subarachnoid space and not subjected to external compression. This has been considered in earlier studies as a finding correlated with the presence of spinal dural pulsation.In this study, patients will be placed in the prone position, and the presence of dural pulsation will be evaluated using ultrasound.

The aim of this study is to evaluate the relationship between the presence of spinal dural pulsation and the clinical and radiological findings in patients diagnosed with lumbar spinal stenosis.

This study has been approved by the Marmara University Faculty of Medicine Non-Pharmaceutical and Non-Medical Device Clinical Trials Ethics Committee with the ethics approval number 09.2025.25-0459.

ELIGIBILITY:
Inclusion criteria

* Aged between 18 and 85 years
* Patients experiencing low back and/or leg pain attributable to lumbar spinal stenosis
* Presence of lumbar spinal stenosis at least at one level consistent with clinical symptoms on lumbar MRI
* Willingness to participate in the study Exclusion criteria
* Body Mass Index (BMI) ≥ 35 kg/m²
* Patients with radiculopathy due to lumbar disc herniation
* Patients with axial low back pain caused by facet syndrome, sacroiliac dysfunction, or discogenic pain
* History of lumbar spine surgery
* Individuals with mental retardation
* Patients with major psychiatric comorbidities
* Patients with congenital spinal anomalies
* Inflammatory rheumatic diseases characterized by osteophyte formation and ligament calcification, such as ankylosing spondylitis and diffuse idiopathic skeletal hyperostosis (DISH)
* Pregnancy
* Patients with heart failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 85 years diagnosed with lumbar spinal stenosis based on physical examination, clinical evaluation, and lumbar magnetic resonance imaging.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The Numeric Rating Scale (NRS) | At the time of data collection
  The Numeric Rating Scale (NRS) is a unidimensional, self-reported measure of pain intensity that is widely used in both clinical practice and research, including studies involving patients with chronic pain. On this scale, patients rate their current level of pain on an 11-point numeric range from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable." Higher scores indicate greater pain intensity.
Oswestry Disability Index | At the time of data collection
  The Oswestry Disability Index (ODI) is a widely used and validated questionnaire designed to assess the degree of disability and functional impairment in patients with low back pain. It evaluates the impact of pain on various aspects of daily living and physical function through ten sections, each scored from 0 to 5, with higher scores indicating greater disability. The total score is converted into a percentage by dividing the obtained score by the maximum possible score and multiplying by 100, yielding a final score ranging from 0% (no disability) to 100% (maximum disability).
SHORT FORM-12 | At the time of data collection
  The Short Form-12 (SF-12) is a health-related quality of life assessment tool that summarizes an individual's physical and mental health status through 12 items. It is a shortened version of the SF-36 questionnaire and measures eight health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The SF-12 produces two composite scores - the Physical Component Summary (PCS) and the Mental Component Summary (MCS) - which are standardized to a mean of 50 and a standard deviation of 10 in the general population. Higher scores indicate better health status and quality of life.
Walking Distance Capacity | At the time of data collection

SECONDARY OUTCOMES:
Dural anteroposterior diameter measured by MRI at the stenotic level | At the time of data collection
Dural cross-sectional area measured by MRI at the stenotic level | At the time of data collection
Schizas classification of the stenotic level on MRI | At the time of data collection
  The Schizas classification is a qualitative grading system used to assess the severity of lumbar spinal canal stenosis on axial T2-weighted magnetic resonance imaging (MRI). It is based on the morphology of the dural sac and the distribution of cerebrospinal fluid (CSF) and nerve rootlets within the canal.
  The classification includes five grades (A-E):
  Grade A: Clearly visible CSF surrounding all cauda equina rootlets (no stenosis).
  Grade B: Some aggregation of rootlets, but CSF still visible (mild stenosis).
  Grade C: Rootlets form a dense bundle with minimal CSF signal (moderate stenosis).
  Grade D: No visible CSF, rootlets fill the dural sac (severe stenosis).
  Grade E: Dural sac completely obliterated or replaced by epidural fat or fibrosis (extreme stenosis).
  Higher grades correspond to more severe central canal stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma B Akdağ, Research Assistant, Principal Investigator — Marmara University Faculty of Medicine ,Marmara University, Department of Physical Medicine and Rehabilitation; Osman H Gündüz, Professor, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine; Serdar Kokar, Associate Professor, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine; Savaş Şencan, Associate Professor, Study Director — Algology Division, Department of Physical Medicine and Rehabilitation, Marmara University Faculty of Medicine
Locations (1):
- Marmara University Faculty of Medicine, Pendik Training and Research Hospital, Algology Department, Pendik, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No